CLINICAL TRIAL: NCT01532128
Title: Effect of BIA 9-1067 on Rasagiline Pharmacokinetics in Healthy Subjects
Brief Title: Effect of BIA 9-1067 on Rasagiline Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-112
Record Dates: First submitted 2012-01-23; First posted 2012-02-14 (Estimated); Results first posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline; opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Period 1: rasagiline 1 mg Period 2: 50 mg BIA 9-1067. 1 hour later rasagiline 1 mg Period 3: rasagiline 1 mg concomitantly with BIA 9-1067 50 mg
  Interventions: Drug: rasagiline; Drug: BIA 9-1067
- Group 2 (Experimental): Period 1: rasagiline 1 mg concomitantly with BIA 9-1067 50 mg Period 2: rasagiline 1 mg Period 3: 50 mg BIA 9-1067. 1 hour later rasagiline 1 mg
  Interventions: Drug: rasagiline; Drug: BIA 9-1067
- Group 3 (Experimental): Period 1: 50 mg BIA 9-1067. 1 hour later rasagiline 1 mg Period 2: rasagiline 1 mg concomitantly with BIA 9-1067 50 mg Period 3: rasagiline 1 mg
  Interventions: Drug: rasagiline; Drug: BIA 9-1067

INTERVENTIONS:
Drug: rasagiline — 1 mg rasagiline (single-dose)
Drug: BIA 9-1067 — 50 mg BIA 9-1067 (single-dose)

SUMMARY:
The purpose of this study is to investigate the effect of BIA 9-1067 on rasagiline pharmacokinetics in healthy subjects.

DETAILED DESCRIPTION:
Single-centre, open-label, randomised, three-way crossover study consisting of 3 single-dose periods separated by a washout of 14 days or more

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were able and willing to give written informed consent.
* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Subjects who had negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening
* Subjects who had clinical laboratory test results clinically acceptable at screening and admission to each treatment period.
* Subjects who had a negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Subjects who were non-smokers or ex-smokers for at least 3 months.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier or intrauterine device.
* (If female) She had a negative pregnancy test (β-HCG) at screening and admission to each treatment period.

Exclusion Criteria:

* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular,psychiatric,musculoskeletal, genitourinary,immunological,dermatological,endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had any significant abnormality in the coagulation tests.
* Subjects who had any significant abnormality in the liver function tests (a case-by-case decision for any abnormality was to be discussed with the Sponsor before inclusion).
* Subjects who had a history of relevant atopy or drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 14 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process at screening or admission to each treatment period.
* Subjects who had acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period.
* Subjects who had received fluoxetine within 5 weeks of admission to the first period.
* Subjects who had used any other medicines within 2 weeks of admission to first period that could affected the safety or other study assessments, in the investigator's opinion.
* Subjects who had previously received BIA 9-1067.
* Subjects who have used any investigational drug or participated in any clinical trial within 90 days prior to screening.
* Subjects who have donated or received any blood or blood products within the 3 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who could not communicated reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an approved effective contraceptive method (double-barrier, intra-uterine device) or she uses oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Béatric Astruc, MD, Principal Investigator — Biotrial - Human Pharmacology Unit
Locations (1):
- BIOTRIAL, Rennes, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 4 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Time Frame: pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Rasagiline Alone: Rasagiline alone.
- Rasagiline 1 h After BIA 9-1067: Rasagiline 1 h after BIA 9-1067.
- Rasagiline Concomitant BIA 9-1067: Rasagiline concomitant BIA 9-1067.
Arm/Group | Rasagiline Alone | Rasagiline 1 h After BIA 9-1067 | Rasagiline Concomitant BIA 9-1067
Number analyzed (Participants) | 24 | 24 | 24
ng/mL
  BIA 9-1067 | NA (NA) — BIA 9-1067 was not administered | 672 (226) | 643 (232)
  Rasagiline | 6152 (2245) | 6.058 (2.399) | 6.078 (2.255)

2. Secondary Outcome: Tmax - Time of Occurrence of Cmax
Time Frame: pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | Rasagiline Alone | Rasagiline 1 h After BIA 9-1067 | Rasagiline Concomitant BIA 9-1067
Number analyzed (Participants) | 24 | 24 | 24
hours
  BIA 9-1067 | NA [NA to NA] — BIA 9-1067 was not administered | 2.00 [1.0 to 4.0] | 2.50 [0.75 to 4.0]
  Rasagiline | 0.50 [0.25 to 1.5] | 0.50 [0.25 to 1.5] | 0.50 [0.25 to 1.5]

3. Secondary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve From Time 0 to Last Observed Concentration
Time Frame: pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Rasagiline Alone | Rasagiline 1 h After BIA 9-1067 | Rasagiline Concomitant BIA 9-1067
Number analyzed (Participants) | 24 | 24 | 24
ng.h/mL
  BIA 9-1067 | NA (NA) — BIA 9-1067 was not administered | 2133 (964.1) | 1980 (861.1)
  Rasagiline | 4.323 (0.9727) | 4.431 (1.010) | 4.391 (0.8782)

ADVERSE EVENTS:
Arm/Group | Before Treatment | Rasagiline Alone | Rasagiline 1 h After BIA 9-1067 | Rasagiline Concomitant BIA 9-1067
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 1/24 | 6/24 | 3/24 | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Before Treatment (N=24) | Rasagiline Alone (N=24) | Rasagiline 1 h After BIA 9-1067 (N=24) | Rasagiline Concomitant BIA 9-1067 (N=24)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 3 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other